CLINICAL TRIAL: NCT06676540
Title: Effect of Eccentric Exercise Training on Spasticity, Walking and Balance in Individuals With Spastic Cerebral Palsy
Brief Title: Effect of Eccentric Exercise on Spasticity, Walking and Balance in Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, HAKAN AYDIN, M.Sc. Pt., Lokman Hekim University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Lokman Hekim Üniversitesi
Record Dates: First submitted 2024-10-13; First posted 2024-11-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy, Spastic
Keywords: Gait Analysis; Postural Balance; Cerebral Palsy; eccentric exercise
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurodevelopmental Therapy (NDT) (Active Comparator): The Neurodevelopmental Therapy (NDT) treatment program, which was determined by the physiotherapist to be individual and suitable for the needs of the cases in both groups participating in the study, will continue throughout the study, with 2 sessions per week and 40 minutes each session. The orthoses and assistive devices used by the cases will continue to be used without any changes and no changes will be made to the treatment program.
  Interventions: Other: Neurodevelopmental Therapy (NDT)
- Neurodevelopmental Therapy (NDT) and Eccentric Exercise Training Group (NDT+EE) (Experimental): The subjects in the study group will be applied NDT 20 minutes twice a week, each session lasting 40 minutes, and in addition, an eccentric exercise program of 20 minutes will be applied in each session. For eccentric exercise training, a functional eccentric exercise program will be applied especially for the hip flexor (m. iliopsoas, m. rectus femoris) muscle group, which is the most common and intense spasticity seen in the lower extremities, hip adductors (m. adductor magnus and minimus, m. adductor longus and brevia, m. pectineus, m. gracillis), knee flexors (m. semitendinosus, m. semimembranouzsu, m. biceps femoris) and plantar flexors (m. gastrocnemius, m. soleus and m. tibialis posterior). If the orthosis used by the individual is applied during the eccentric exercise program, it will be removed.
  Interventions: Other: Neurodevelopmental Therapy (NDT) and Eccentric Exercise Training Group (NDT+EE); Other: Neurodevelopmental Therapy (NDT)

INTERVENTIONS:
Other: Neurodevelopmental Therapy (NDT) and Eccentric Exercise Training Group (NDT+EE) — Including Functional Eccentric Exercises Applied to Individuals with Cerebral Palsy
  Arms: Neurodevelopmental Therapy (NDT) and Eccentric Exercise Training Group (NDT+EE)
Other: Neurodevelopmental Therapy (NDT) — This application includes rehabilitation methods frequently used in pediatric rehabilitation.

SUMMARY:
Our clinical research study is planned as a randomized controlled study and will use a stratified randomization method. The aim of this study is to investigate the effects of eccentric exercise training on spasticity, walking and balance in individuals with spastic Cerebral Palsy (CP). Individuals with spastic unilateral SP (hemiparetic) and bilateral SP (diparetic) diagnosis, Gross Motor Function Classification System (GMFCS) Level I, II and III, aged between 6-18 years will be included in the study.

DETAILED DESCRIPTION:
As a result of the G-power analysis, it was revealed that a total of 42 individuals should be included in the control and study groups. In our study, a control group of 21 people (Neurodevelopmental Treatment Group-NGT/2 days per week, 40 minutes) and an experimental group (Neurodevelopmental Treatment + Eccentric Exercise Group-NGT+EE/2 sessions per week, 20 minutes NGT + 30 minutes eccentric exercise program) will be formed. After the initial evaluations, 2 physiotherapy sessions per week will be applied to both groups for 8 weeks and then the final evaluations will be made and the obtained data will be compared with the initial evaluation data to reveal the statistical effect of eccentric exercises on spasticity, walking and balance parameters.

The hypotheses of the study are as follows:

H1: Eccentric exercise training for spastic lower extremity muscles in individuals with spastic cerebral palsy has an effect on spasticity severity.

H2: Eccentric exercise training for spastic lower extremity muscles in individuals with spastic cerebral palsy has an effect on gait parameters.

H3: Eccentric exercise training for spastic lower extremity muscles in individuals with spastic cerebral palsy has an effect on balance parameters.

H4: Eccentric exercise training for spastic lower extremity muscles in individuals with spastic cerebral palsy has an effect on quality of life, activities of daily living (ADL), and participation.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 6-18 and diagnosed with spastic hemiparetic or spastic diparetic CP,
* Being at level I, II or III according to GMFCS,
* Having increased muscle tone in hip flexor, hip adductor, knee flexor, knee extensor or ankle plantar flexor muscles according to MTS,
* Giving informed consent including detailed information prepared for the study (by parent/guardian).

Exclusion Criteria:

* Having received botox or surgery in the last 6 months.
* Not signing the consent form.
* Having limited cooperation regarding perception or performance of exercises required for the study.
* Having a systemic disease in addition to CP.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Functional Balance | 2 month
  Functional Balance will be evaluated with the 'Pediatric Balance Scale (PBS)'. PBS has been reported to be valid and reliable in the assessment of functional balance in patients with CP. This scale evaluates many different situations that will challenge balance during position transitions and upright positions during daily living activities. It consists of 14 questions that include activities such as sitting to standing, standing, transfers, taking steps, standing on one leg, turning, bending, and reaching. Each question is scored between 0-4. The total score of the test is 56. High scores indicate good balance performance.
Stabilometric Balance Assessment (eyes open and eyes closed balance) | 2 month
  In this assessment, which is performed while standing still on a pedobarographic analysis device, objective data on postural sway and balance can be obtained together with static plantar pressure data. The data obtained with eyes open and closed are recorded. The decrease in postural sway between the two measurements with the numerical data obtained indicates that balance is better.
Visual Gait Analysis | 2 month
  Will be evaluated with Edinburgh Visual Gait Analysis (EVGA). EVGA was developed to create an easy-to-use gait score that is compatible with 3-D gait analyses in children with CP. EGGA is a valid and reliable method for use in children with CP. EVGA consists of 17 items scored separately for the right and left lower extremities. The assessments include 6 anatomical levels: trunk, pelvis, hip, knee, ankle, and foot. These anatomical levels are assessed in the sagittal, coronal, and transverse planes. A 3-point ordinal scale is used for scoring. A score of 0 indicates normal, a score of 1 indicates moderate deviation from normal, and a score of 2 indicates significant deviation from normal. The scores obtained by watching camera recordings for each lower extremity are added up and a single score is obtained. A low score indicates normal; a high score indicates abnormal gait.
Muscle Tone | 2 month
  Will be evaluated with 'Modified Ashworth Scale (MAS)'. It is a measurement method based on determining the resistance shown by the spastic muscle during passive movement of the relevant extremity. The 5-degree MAS was obtained by adding the value 1+ to the Asworth scale, which evaluates muscle tone between 0 and 4. The value 0 indicates a normal situation where there is no increase in muscle tone; while the value 4 indicates the maximum increase in muscle tone.
Spasticity | 2 month
  Will be evaluated with 'Modified Tardieu Scale (MTS)'. Tardieu Scale was developed in 1954 and is a scale that evaluates spasticity with passive movement. The evaluation is made at the rate of the extremity segments falling with gravity, slower than this rate (R2) and faster than this rate (R1). This scale has been modified to evaluate at two different speeds, R1 and R2. For R1 and R2 values, the points where the muscle first resists during joint movement are measured with a goniometer. In the R1 evaluation, the sense of catching caused by the increased stretch reflex in fast joint movement (spasticity) is evaluated, while in the R2 evaluation, information is obtained about the range of motion and muscle length in slow joint movement. According to the MTS, it is accepted that the severity of spasticity increases as the difference between the R1 and R2 values increases.

SECONDARY OUTCOMES:
Lower extremity Range of Motion | 2 month
  Lower extremity active and passive normal joint range of motion values will be measured in degrees with a standard universal goniometer.
Boyd and Graham's Selective Motor Control (SMC) Test | 2 month
  The "Selective Motor Control of Dorsiflexion Test" or "Boyd and Graham's Selective Motor Control (SMC) Test", defined by Boyd and Graham, was developed to evaluate ankle dorsiflexion (DF) SMC. It is associated with foot functions observed during walking. It is scored between 0 and 4. The person sits tall with hip flexion and knee extension so that they can see their feet and is asked to dorsiflex. A value of 0 indicates that there is no active ankle DF. A value of 4 indicates that isolated DF is performed without hip and knee flexion. A high score indicates that selectivity is good.

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No